CLINICAL TRIAL: NCT06612593
Title: The Effect of Cilostazol on the Clinical Outcome of Patients with Parkinson's Disease
Brief Title: Cilostazol in Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doha Adel, Clinical Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHDIRB2020110301 REC # 282
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Parkinson's Disease
Keywords: PD, Parkinson's Disease, Cilostazol, Neuroinflammation, Oxidative Stress, Anti-inflammatory, Anti-oxidant, Neuroprotective, MDS-UPDRS
MeSH Terms: conditions — Parkinson Disease; Neuroinflammatory Diseases | interventions — Cilostazol

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Single-blinded Controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cilostazol Group (Experimental): 25 participants will receive the standard treatment and cilostazol at a dose of 50 mg twice daily for a month, then the dose will be increased to 100 mg twice daily for 5 months.
  Interventions: Drug: Cilostazol; Drug: Standard treatment
- Control Group (Active Comparator): 25 participants will receive the standard treatment and the placebo twice daily for 6 months.
  Interventions: Drug: Placebo; Drug: Standard treatment

INTERVENTIONS:
Drug: Cilostazol — 2 tablets of 50 mg cilostazol will be received for 4 weeks, then the does will be 2 tablets of 100 mg cilostazol twice daily for 20 weeks
  Arms: Cilostazol Group
Drug: Placebo — The patient will receive 2 tablets twice daily
  Arms: Control Group
Drug: Standard treatment — It includes Levodopa with a dose of 375 to 1000mg daily and Dopamine agonists with a dose of 1.5 to 5 mg daily.

SUMMARY:
Parkinson's disease is the second most common neurodegenerative diseases. The conventional treatment for PD has included dopaminergic treatment as Levodopa\carbidopa or dopamine agonists, anti-cholinergics, MAOI, catechol-o-methyl transferase (COMT) inhibitors, and amantadine. Although these options have been found to be effective, they could only improve the disease symptoms, but do not modify the disease progression. Hence, researchers have focused on developing disease-modifying agents to stop or slow the progression acting as neuroprotective agents. Since the inflammation and oxidative stress play an important role in the pathophysiologic progression of PD, recent studies have investigated the mitigation of the disease pathology through anti-inflammatory and anti-oxidant agents.

Cilostazol has been found to have anti-inflammatory, antioxidant, and neuroprotective effect, and has been evaluated through two animal studies to prove that it possess these effects through dampening NF-κB, and its downstream effectors including TNF-α and IL-1β, reversing the activation of glycogen synthase kinase-3 β (GSK-3β), a pivotal effector in neuronal apoptosis, contributing in preserving dopaminergic neuron integrity clarifying the enhance motor activity, activating nuclear factor erythroid-related factor 2/ heme oxygenase 1 (Nrf2/HO-1), suppressing High mobility group box 1 protein/Toll-like receptor 4 (HMGB1/TLR4) axis, and upregulatig Phosphoinositide 3-kinases/ Protein kinase B (PI3K/Akt) besides mammalian target of rapamycin (mTOR) inhibition. Hence, Cilostazol might be a potential candidate to improve the clinical outcome in PD patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease, affecting about 1% of the elderly population, with 5 to over 35 new cases in 100,000 per year diagnosed with PD, with a prevalence of over 10 million people worldwide. This number is projected to increase to more than 12 million by 2040. The incidence of PD increase with age but it can affect people less than 50 years old. In the Eastern Mediterranean Region (EMR), the prevalence rate of PD increased by 42.3% over the period 1990-2016, and reached 87.1 per 100,000 in 2016. Factors that cause PD are multifactorial including genetic predispositions, environmental toxins, and aging leading to disease initiation and progression.

Parkinson's disease is a chronic condition characterized by the slow progression of the dopaminergic neuronal degeneration with irreversible loss of dopamine (DA). It is associated with motor symptoms as bradykinesia, resting tremor, rigidity, and postural instability. It also affects other extra-nigral dopaminergic, cholinergic and serotoninergic tracts, leading to non-motor symptoms as anosmia, sleep disorders and constipation as well as cognitive and psychiatric symptoms like cognitive impairment, dementia and depression.

Cognitive decline is a common non-motor symptom in PD, and an important source of patient disability and caregiver burden. The pathophysiology of cognitive impairment in PD is complex and likely involves a disruption of several distinct neuronal networks occurring over time. The timing, profile and rate of cognitive decline vary widely among individuals with PD and can range from normal cognition to mild cognitive impairment and dementia.

The pathogenesis of PD is not fully understood, however, several studies have revealed that the inflammation, oxidative stress, and neuronal apoptosis have a major role in its progression. In addition, PD was found to be linked with the reduction of the regional cerebral blood flow (rCBF). This reduced cerebral blood flow has been found to be associated with the occurrence of cognitive impairment and dementia.

Neuroinflammation in PD has been evidenced through several human and animal studies. It may result from the consequences of ongoing neuronal cell death in PD, the aggregation of misfolded α-Synuclein, microgliosis and astrogliosis, peripheral inflammation and PD-risk-associated genes. Any of these factors will result in the activation of microglia, CNS-resident macrophages important for normal CNS functioning, and production of pro-inflammatory mediators as cytokines (IL1, IL6, and TNFα) chemokines and reactive oxygen species, leading to the exacerbation of DA neuron degeneration.

In addition, PD has been linked to decreased levels of brain-derived neurotrophic factor (BDNF). Brain-derived neurotrophic factor belongs to a family of proteins called neurotrophin family of growth factors, that support differentiation, maturation, and survival of neurons in the nervous system and shows a neuroprotective effect under adverse conditions, such as glutamatergic stimulation, cerebral ischemia, hypoglycemia, and neurotoxicity. Studies has investigated the reduced expression of BDNF through the decreased levels of BDNF in the substantia nigra pars compacta in post-mortem brain tissues, and decreased serum levels of BDNF in PD patients. These reduced levels of BDNF have been attributed to the inflammation and neurodegeneration.

Oxidative stress along with inflammation has been evidenced to play a critical role in the dopaminergic neuronal degeneration. The sources and mechanisms for generation of reactive oxygen species (ROS) include dopamine metabolism, mitochondrial dysfunction, iron, neuroinflammation, calcium, and aging. Additionally, cellular homeostatic processes including the ubiquitin-proteasome system, the main pathway through which cells degrade and remove damaged and unwanted proteins, and mitophagy are affected by oxidative stress. Together, these various mechanisms contributes to the neurodegeneration in PD where primary insults lead to oxidative stress, which damages key cellular proteins and the disruption of lipid membranes causing more ROS production. The role of oxidative stress is supported by postmortem brain analyses showing increased levels of 4-hydroxyl-2-nonenal (HNE), a by-product of lipid peroxidation, and DNA and RNA oxidation products 8-hydroxy-deoxyguanosine and 8-hydroxy-guanosine. In addition, oxidative stress has been found to be involved in the pathway leading to apoptotic cell death which has been investigated through research studies involving human and animal PD models.

In addition, neuroinflammation and oxidative stress have been found to contribute to the development of cognitive impairment in PD patients.

For many years, the conventional treatment for PD has included dopaminergic treatment as Levodopa\carbidopa or dopamine agonists, anti-cholinergics, MAOI, catechol-o-methyl transferase (COMT) inhibitors, and amantadine. Although these options have been found to be effective, they could only improve the disease symptoms, but do not modify the disease progression. Hence, researchers have focused on developing disease-modifying agents to stop or slow the progression acting as neuroprotective agents. Since the inflammation and oxidative stress play an important role in the pathophysiologic progression of PD, recent studies have investigated the mitigation of the disease pathology through anti-inflammatory and anti-oxidant agents. Human and animal studies have found that the anti-inflammatory agents protect dopaminergic neurons and ameliorate the disease associated symptoms. Several anti-oxidant agents, such as curcumin and vitamin E, have been investigated in PD patients. These agents have shown an effect on reducing dopamine oxidation, delaying the disease progression, and reducing the motor deficit. Therefore, more treatment options attempting to stop the pathophysiologic alterations should be explored.

Cilostazol (CSZ), a 2-oxo-quinoline derivative, is a selective inhibitor of phosphodiesterase-3 that increases intracellular cAMP levels and activates protein kinase A. Cilostazol is a lipophilic drug that can cross the blood brain barrier, with anti-platelet, anti-mitogenic, and vasodilating properties, and is FDA approved for the treatment of ischemic symptoms of peripheral vascular diseases, including intermittent claudication, and the prevention of cerebral and myocardial infarction. In addition, cilostazol improves the cerebral blood flow and cerebral function during the chronic stage of cerebral infarction. Recently, it has noteworthy antioxidant, anti-inflammatory, and anti-apoptotic properties.

Cilostazol has shown potent anti-inflammatory action through inhibiting toll-like receptor (TLR) signaling-mediated NF-κB activation and the production of pro-inflammatory cytokine as IL-6, prostaglandin E2, interleukin-1 (IL-1), tumor necrosis factor (TNF-α), and monocyte chemo-attractant protein-1 (MCP-1). It can also exert its antioxidant effects through reversing the GSH depletion, normalizing hippocampal oxidative stress biomarkers as Glutathione peroxidase and superoxide dismutase, and reducing the MDA levels. Several studies have demonstrated that cilostazol has neurotrophic effect through improving the expression of neurotrophic factors, and in turn, it increases the levels of BDNF.

Cilostazol has been used in experimental studies for several neurodegenerative disorders as Parkinson's disease, Huntington disease, and Alzheimer's disease (AD) for its neuroprotective effect due to its neuroprotective effect. This neuroprotective effect has been demonstrated through maintaining the brain function in animal models with focal cerebral ischemia attributed to its anti-apoptotic properties, and preventing the hypoperfusion-induced cognitive impairment in animal models with vascular dementia. In addition, it has beneficial effects on cognitive and regional cerebral blood flow (rCBF) deficits in the elderly patients, and is associated with a decreased risk of dementia, and slowing the rate of cognitive decline on the MMSE in mild cognitive impairment patients, mild dementia patients, and Alzheimer's disease patients. From the previously mentioned data, cilostazol can act as a potential candidate for PD patients.

Cilostazol has been evaluated in 2 animal studies and it was found that cilostazol possessed an anti-inflammatory, anti-oxidant, and anti-apoptotic effects in PD through dampening NF-κB, and its downstream effectors including TNF-α and IL-1β, reversing the activation of glycogen synthase kinase-3 β (GSK-3β), a pivotal effector in neuronal apoptosis, contributes preserving dopaminergic neuron integrity clarifying the enhanced motor activity, activating nuclear factor erythroid-related factor 2/ heme oxygenase 1 (Nrf2/HO-1), suppressing High mobility group box 1 protein/Toll-like receptor 4 (HMGB1/TLR4) axis, and upregulatig Phosphoinositide 3-kinases/ Protein kinase B (PI3K/Akt) besides mammalian target of rapamycin (mTOR) inhibition.

Cilostazol has a good safety profile beside its potent anti-inflammatory and antioxidant effects, which make it a candidate for many experimental and clinical trials. Its more common side effects include headache (27-34%) and GI symptoms (12-19%). It has other side effects as ecchymoses, anemia, edema, dizziness, palpitations, rhinitis, pharyngitis, chest pain, allergy, myalgia, and sleep disturbance, but they are less common (<2%).

ELIGIBILITY:
Inclusion Criteria:

* -Adult patients.
* Both males and females will be included
* Diagnosed Parkinson's disease according to the MDS criteria 2015
* At least 5 years of disease duration
* On stable Levodopa\carbidopa regimen for the past 6 months.
* Clinically diagnosed with dyskinesia

Exclusion Criteria:

* -Secondary causes of Parkinsonism
* Atypical parkinsonian syndromes
* Active malignancy
* Known intolerance or hypersensitivity to cilostazol
* Participation in other interventional trials
* Patients with hepatic (AST and ALT more than 3 times the upper normal limit) or renal impairment (eGFR less than 60 ml\min).
* Patients receiving warfarin, other anti-coagulants or anti-platelet therapy.
* Patients with Congestive heart failure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the severity of Parkinson's disease symptoms using the Movement Disorder Society-unified Parkinson's disease rating scale (MDS-UPDRS)Assessment | 6 months
  MDS-UPDRS will be performed at baseline, after 12weeks and after 24 weeks. MDS-UPDRS, the revised form of UPDRS, is the most common tool used to measure progression in PD patients. It consists of 4-subscale structure: Part I, Non-Motor Aspects of Experiences of Daily Living (13 items); Part II, Motor Aspects of Experiences of Daily Living (13 items); Part III, Motor Examination (33 items); and Part IV, Motor Complications (6 items). The scores in each item vary from 0 (normal) to 4(severe).

SECONDARY OUTCOMES:
Serum Level of BDNF Assessment: | 6 months
  Blood sample will be withdrawn from each patient at baseline and after 24 weeks. Samples will be centrifuged, and the sera will be separated and stored at -80C till analysis. Serum BDNF will be measured using human BDNF ELISA kit at baseline and after 24 weeks.
Safety Assessment | 6 months
  Side effects include headache, ecchymoses, edema, dizziness, palpitations, rhinitis, pharyngitis, chest pain, allergy, myalgia, and sleep disturbance. All subjects will be educated about the adverse effects of cilostazol and will be required to report the occurrence of any of them. Patients will be followed up every 2 weeks by phone call and every month during clinic visits to check for the occurrence of any side effects.
Assessment of the degree of cognitive impairment with The Montreal Cognitive Assessment (MoCA) | 6 months
  Assessment of cognitive impairment is performed at baseline, after 12 weeks and after 24 weeks using the MoCA test. The MoCA test is a one-page 30-point test administered in 10 minutes as a rapid screening instrument for CI. It consists of 6 domains: The short-term memory recall task (5 points) ; Visuospatial abilities (4points) ; Executive functions (4 points); Attention, concentration, and working memory (6 points); Language (5 points) ; orientation to time and place (6 points). The total possible score is 30 points; a score of 26 or above is considered normal.
Assessment of Quality of life (QoL) USING the PDQ-39 questionnaire | 6 months
  Assessment of QOL will be performed at baseline, after 12 weeks and after 24 weeks using the PDQ-39 questionnaire. The PDQ-39 questionnaire is considered as the most appropriate instrument to evaluate QoL in PD patients. It consists of 39 multiple-choice questions items in eight domains: Mobility (10 items); Activities of Daily Living ADL (6 items); Emotional well-being (6 items); Stigma (4 items); Social support (3 items); Cognition (4items); Communication (3 items); and Bodily discomfort (3 items) ", with five possible answers: "Never"; "Occasionally"; "Sometimes"; "Often"; "Always" or "Cannot do at all". Each individual's total score is calculated as follows:
  100 x (The sum of the patient's score in the 39 questions /4 x 39) he total score varies from 0 indicating the least impact on QoL (no problem); to 100 indicating the maximum impact on QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdallah MS, Ramadan AN, Omara-Reda H, Mansour NO, Elsokary MA, Elsawah HK, Zaki SA, Abo Mansour HE, Mosalam EM. Double-blind, randomized, placebo-controlled pilot study of the phosphodiesterase-3 inhibitor cilostazol as an adjunctive to antidepressants in patients with major depressive disorder. CNS Neurosci Ther. 2021 Dec;27(12):1540-1548. doi: 10.1111/cns.13731. Epub 2021 Sep 21. PMID 34545997
- [Background] Arai H, Takahashi T. A combination therapy of donepezil and cilostazol for patients with moderate Alzheimer disease: pilot follow-up study. Am J Geriatr Psychiatry. 2009 Apr;17(4):353-4. doi: 10.1097/JGP.0b013e31819431ea. No abstract available. PMID 19307864
- [Background] Holden SK, Finseth T, Sillau SH, Berman BD. Progression of MDS-UPDRS Scores Over Five Years in De Novo Parkinson Disease from the Parkinson's Progression Markers Initiative Cohort. Mov Disord Clin Pract. 2018 Jan-Feb;5(1):47-53. doi: 10.1002/mdc3.12553. Epub 2017 Sep 22. PMID 29662921
- [Background] Parkinson Study Group. Effects of tocopherol and deprenyl on the progression of disability in early Parkinson's disease. N Engl J Med. 1993 Jan 21;328(3):176-83. doi: 10.1056/NEJM199301213280305. PMID 8417384
- [Background] Hedya SA, Safar MM, Bahgat AK. Cilostazol Mediated Nurr1 and Autophagy Enhancement: Neuroprotective Activity in Rat Rotenone PD Model. Mol Neurobiol. 2018 Sep;55(9):7579-7587. doi: 10.1007/s12035-018-0923-1. Epub 2018 Feb 10. PMID 29429051
- [Background] Howells DW, Porritt MJ, Wong JY, Batchelor PE, Kalnins R, Hughes AJ, Donnan GA. Reduced BDNF mRNA expression in the Parkinson's disease substantia nigra. Exp Neurol. 2000 Nov;166(1):127-35. doi: 10.1006/exnr.2000.7483. PMID 11031089
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Rahman TT, El Gaafary MM. Montreal Cognitive Assessment Arabic version: reliability and validity prevalence of mild cognitive impairment among elderly attending geriatric clubs in Cairo. Geriatr Gerontol Int. 2009 Mar;9(1):54-61. doi: 10.1111/j.1447-0594.2008.00509.x. PMID 19260980
- [Background] Safiri S, Noori M, Nejadghaderi SA, Mousavi SE, Sullman MJM, Araj-Khodaei M, Singh K, Kolahi AA, Gharagozli K. The burden of Parkinson's disease in the Middle East and North Africa region, 1990-2019: results from the global burden of disease study 2019. BMC Public Health. 2023 Jan 16;23(1):107. doi: 10.1186/s12889-023-15018-x. PMID 36642724
- [Background] Sakamoto T, Ohashi W, Tomita K, Hattori K, Matsuda N, Hattori Y. Anti-inflammatory properties of cilostazol: Its interruption of DNA binding activity of NF-kappaB from the Toll-like receptor signaling pathways. Int Immunopharmacol. 2018 Sep;62:120-131. doi: 10.1016/j.intimp.2018.06.021. Epub 2018 Jul 10. PMID 30005227